CLINICAL TRIAL: NCT06445881
Title: A Multi-center, Prospective, Exploratory Study Evaluating the Efficacy and Safety of a Modified Si Jun Zi Tang Formula in the Perioperative Treatment of Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Modified Si Jun Zi Tang in Perioperative NSCLC Treatment
Acronym: MSJZT-NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240018C-R1
Record Dates: First submitted 2024-06-02; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer; Perioperative Complication
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Si Jun Zi Tang Combined with Chemotherapy and Immunotherapy (Experimental): Participants will receive Modified Si Jun Zi Tang combined with chemotherapy (albumin-bound paclitaxel or pemetrexed + carboplatin) and PD1 monoclonal antibody, followed by surgery if feasible. Postoperatively, they will continue with Modified Si Jun Zi Tang and PD1 monoclonal antibody for up to one year.
  Interventions: Drug: Modified Si Jun Zi Tang
- Standard Chemotherapy and Immunotherapy (No Intervention): Participants will receive standard chemotherapy (albumin-bound paclitaxel or pemetrexed + carboplatin) and PD1 monoclonal antibody, followed by surgery if feasible. Postoperatively, they will continue with PD1 monoclonal antibody for up to one year.

INTERVENTIONS:
Drug: Modified Si Jun Zi Tang — Modified Si Jun Zi Tang is a classic formula in traditional Chinese medicine, known for its benefits in unifying and strengthening the spleen.
  Arms: Modified Si Jun Zi Tang Combined with Chemotherapy and Immunotherapy

SUMMARY:
Chemotherapy combined with immunotherapy is the current standard perioperative treatment for non-small cell lung cancer (NSCLC). However, this regimen has multiple side effects and shows variable efficacy among individuals. In China, adjunctive traditional Chinese medicine is widely accepted by lung cancer patients. Modified Si Jun Zi Tang, a classic formula in traditional Chinese medicine, is known for its benefits in unifying and strengthening the spleen. This study aims to evaluate whether the addition of Modified Si Jun Zi Tang to chemotherapy and immunotherapy during the neoadjuvant phase can improve the R0 resection rate, objective response rate (ORR), and safety in patients with resectable and potentially resectable NSCLC. Secondary objectives include assessing whether this combination can improve 1-year and 2-year disease-free survival (DFS) post-surgery. Additionally, we will collect relevant biological samples to identify tumor markers associated with efficacy, prognosis, and side effects, providing a theoretical basis for modernizing and standardizing traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Pathologically confirmed non-small cell lung cancer (NSCLC) with no prior treatment for this tumor.
3. Clinical stage II-IIIB (N2) tumors assessed as resectable or potentially resectable by a multidisciplinary team (MDT).
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 - 1.
5. Adequate organ function, including:

   Bone marrow: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 80 x 10^9/L, hemoglobin ≥ 90 g/L.

   Liver: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤ 3 times ULN.

   Kidneys: Creatinine clearance rate ≥ 45 mL/min (using the standard Cockcroft-Gault formula) or ≤ 1.5 times ULN.
6. At least one measurable lesion according to RECIST v1.1 criteria.
7. For women: Must be surgically sterilized, postmenopausal, or use highly effective contraception during and for 3 months after treatment; must not be pregnant or breastfeeding during the treatment period.
8. Patients must have compliance and geographic proximity to ensure adequate follow-up.

Exclusion Criteria:

1. Patients with a history of autoimmune diseases, active tuberculosis, active hepatitis (HBV DNA <2000 IU), or HIV infection.
2. Patients expected to be unable to tolerate surgery, such as those with severe cardiopulmonary insufficiency or coagulation disorders (APTT <1.5 times ULN, INR >2.0, PT >16 seconds).
3. History of other malignancies within the past 2 years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin, superficial bladder cancer [Ta, Tis & T1], or papillary thyroid carcinoma.
4. Any unstable systemic disease (including active systemic infections requiring systemic treatment, liver disease, kidney disease, or metabolic disorders, acute cerebral infarction or cerebral hemorrhage, etc.).
5. Significant cardiovascular events: congestive heart failure > NYHA Class 2; unstable angina, active coronary artery disease (CAD) (myocardial infarction over 1 year before study entry is allowed); severe arrhythmias requiring treatment (use of beta-blockers or digoxin is allowed) or uncontrolled hypertension.
6. Significant neurological or psychiatric disorders, including epilepsy, dementia, etc.
7. Patients with interstitial lung disease or a history of interstitial pneumonia.
8. Participation in other anti-tumor drug clinical trials within 4 weeks prior to enrollment.
9. Previous use of PD-1/PD-L1 inhibitors or other anti-tumor immunotherapy drugs.
10. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or planned transplantation.
11. Known allergy to the drugs or drug excipients used in the study or severe allergic reactions to other monoclonal antibodies.
12. Presence of other severe physical or laboratory abnormalities that may increase the risk of participating in the study, interfere with study results, or any other condition that, in the investigator's judgment, may affect the conduct or results of the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | Assessed at the time of surgery, approximately 2-4 months after starting treatment.
  The proportion of patients achieving complete surgical resection with negative margins (R0 resection) after neoadjuvant therapy.
Objective Response Rate (ORR) | Assessed after 2 cycles of treatment (approximately 6 weeks) and before surgery, if applicable.
  The proportion of patients achieving partial or complete response as defined by RECIST v1.1 criteria.
Incidence of Adverse Reactions | Assessed throughout the treatment period, from the start of treatment up to one year post-surgery.
  The proportion of patients experiencing treatment-related adverse reactions, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
1-Year Disease-Free Survival (DFS) | Assessed one year post-surgery.
  The proportion of patients who remain free of disease recurrence or progression one year after surgery.
2-Year Disease-Free Survival (DFS) | Assessed two years post-surgery.
  The proportion of patients who remain free of disease recurrence or progression two years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhen Shan, MD, Principal Investigator — the First Affiliated Hospital of Zhejiang Universtiy
Locations (1):
- the First Affilated Hospital of Zhejiang University, Hangzhou, Zhejiang, China